CLINICAL TRIAL: NCT02317549
Title: Treatment of Septic Shock by Inhibiting Autodigestion and Preserving Gut Integrity With Enteric LB1148 (SSAIL Trial)
Brief Title: Treatment of Septic Shock by Inhibiting Autodigestion and Preserving Gut Integrity With Enteric LB1148
Acronym: SSAIL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inability to enroll
Sponsor: Leading BioSciences, Inc (Industry)
Responsible Party: Sponsor
Organization: Palisade Bio (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LBS-SS201
Record Dates: First submitted 2014-12-11; First posted 2014-12-16 (Estimated); Results first posted 2017-11-20 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Septic Shock
Keywords: sepsis; septic shock; vasodilatory shock; circulatory shock; Systemic Inflammatory Response Syndrome; SIRS; infection; toxemia; gut barrier breakdown; autodigestion; multiorgan failure; MOF; multiorgain dysfunction syndrome; MODS; hyperlactatemia; tissue hypoxia
MeSH Terms: conditions — Shock, Septic; Sepsis; Shock; Systemic Inflammatory Response Syndrome; Infections; Toxemia; Multiple Organ Failure; Hyperlactatemia | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tranexemic Acid (Experimental): Daily a total of 700 mL of LB1148 solution containing 7.5 g of tranexemic acid will be administered orally or via NG/OG/NJ/ND/PEG tube
  Interventions: Drug: LB1148
- Placebo (Placebo Comparator): Daily a total of 700 mL of Placebo solution will be administered orally or via NG/OG/NJ/ND/PEG tube
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LB1148
  Other Names: Tranexamic Acid
  Arms: Tranexemic Acid
Drug: Placebo
  Arms: Placebo

SUMMARY:
Septic shock is a potentially life-threatening condition that can result in multi-organ dysfunction syndrome (MODS) and mortality. LB1148 was formulated to preserve gut integrity during physiological shock and ameliorate the subsequent autodigestion leading to MODS and mortality. The purpose of this study in septic shock patients is to determine if enteral administration of LB1148 will increase the number of days alive without cardiovascular, pulmonary or renal replacement therapy through Day 28.

DETAILED DESCRIPTION:
Primary Objective(s):

The primary objective of this study is to determine if enteral administration of LB1148 will increase the number of days alive without cardiovascular, renal or pulmonary organ support through Day 28.

The secondary objectives of this study are to determine if LB1148 will:

* Reduce mortality at Day 7, Day 28 and Day 90;
* Reduce the number of days to organ dysfunction resolution as evidenced by Sequential Organ Failure Assessment (SOFA) score ≤2 in patients alive on Day 28;
* Reduce the daily organ dysfunction as evidenced by average SOFA score through Day 14 and Day 28;
* Reduce the number of patients with new-onset organ dysfunction at Day 8;
* Increase the number of days alive and free from renal replacement therapy through Day 28;
* Increase the number of days alive and free from renal dysfunction through Day 28;
* Increase the number of days alive and ventilator free through Day 28;
* Increase the number of days alive and free of vasopressors through Day 14 and Day 28;
* Increase the numbers of days alive and free from liver dysfunction through Day 28;
* Increase the number of days alive and not in the Intensive Care Unit (ICU) through Day 28;
* Increase the number of days alive and not in the hospital through Day 28, and
* Improve patient functional outcomes through Day 28 as evidenced by the EuroQoL EQ 5D questionnaire.

In addition, the study will assess the safety and tolerability of LB1148 in patients with septic shock.

The exploratory objectives of this study are to determine if LB1148 will:

* Reduce the number of patients with new-onset organ dysfunction from Day 9 through Day 16;
* Decrease the number of days to normalize serum lactate (≤2.2 mmol/L) through Day 28;
* Reduce the average daily serum lactate levels through Day 8;
* Increase the number of days alive and free from ileus through Day 8 and Day 28.

ELIGIBILITY:
Inclusion Criteria:

1. First episode (during the current hospitalization) of documented or suspected sepsis of peritoneum/abdomen, soft tissue, blood, or non-hospital acquired lung origin.
2. Must be receiving antimicrobial therapy for documented or suspected infection.
3. Must have septic shock requiring vasopressors despite adequate fluid resuscitation of 30 mL/kg crystalloid or colloid equivalent, for either an SBP ≤90 mmHg or a MAP ≤65 mmHg (i.e. must have been unable to maintain adequate blood pressure despite adequate fluid resuscitation without the use of vasopressors). Note: 30 mL/kg crystalloid is equivalent to 15 mL/kg colloids.
4. Must have a requirement for vasopressor support after adequate fluid resuscitation, and, at randomization, must require a minimum dose of at least 1 of the following vasopressors:

   * Norepinephrine ≥5 µg/min;
   * Dopamine ≥10 µg/kg/min;
   * Phenylephrine ≥25 µg/min;
   * Epinephrine ≥5 µg/min, or
   * Vasopressin ≥0.03 units/min.

Exclusion Criteria

Patients will not be eligible for participation in the study if they meet ANY of the following criteria:

1. Age <18 or age ≥76 years.
2. Time elapsed since onset of shock is >24 hours. Onset of shock is defined as the first administration of a vasopressor given by continuous infusion (i.e. not a single bolus of norepinephrine, phenylephrine, or ephedrine).
3. Septic shock episode is the second or greater episode in current hospitalization.

   Note: patients transferred from another healthcare facility that are still within the first 24 hours of the first episode of shock are eligible.
4. Have hospital acquired pneumonia.
5. Have genitourinary infections as the cause of septic shock.
6. Unable to maintain a minimum MAP of 60 mmHg despite the presence of vasopressors and IV fluids.

   Note: brief transient BPs below 60 mmHg are not disqualifying.
7. Have a serum lactate measurement <2.5 mmol/L after adequate fluid resuscitation (refer to Inclusion Criteria #3).
8. Not expected to survive for at least 28 days due to a preexisting, non-shock related medical condition.
9. Highest total SOFA score (known to staff at the time of randomization) during the screening period <6.

   Note: each individual organ component sub-score is calculated from the highest (worst) score obtained for that organ during the screening period, up until randomization.
10. Highest total SOFA score (known to staff at the time of randomization) during the screening period >18.

    Note: each individual organ component sub-score is calculated from the highest (worst) score obtained for that organ during the screening period.
11. Lack of commitment to aggressive source control of infection.
12. The patient or patient's surrogate fails to voluntarily sign an informed consent form (ICF).
13. Ineligible for feeding tube placement.
14. Chronic renal insufficiency requiring hemodialysis not associated with the current episode of sepsis.
15. Chronic pulmonary dysfunction requiring mechanical ventilation unrelated to the current episode of sepsis.
16. Undergoing active radiation or cytotoxic chemotherapy treatment for uncontrolled malignancy.

    Note: hormonal and surgical therapies are permitted.
17. Presence of third degree burns involving >20% body surface area in the 7 days prior to study entry.
18. Known inability to take the study medication (i.e. complete small bowel obstruction).
19. Has acute meningitis.
20. Have any of the following medical conditions:

    * HIV-positive patients whose most recent CD4 count was ≤50/mm3;
    * Neutrophils <1000/mm3 unless due to sepsis;
    * Received chest compressions as part of CPR during this hospitalization without neurologic recovery;
    * Poorly controlled neoplasm;
    * End-stage lung disease or Cystic Fibrosis;
    * End-stage liver disease (Child-Pugh Class C [score >10], evidence of portal hypertension or esophageal varices);
    * Severe congestive heart failure (New York Heart Association [NYHA] Class IV or pre-sepsis ejection fraction <30%);
    * Undergone organ transplant (including bone marrow, heart, lung, liver, pancreas, or small bowel transplantation), or
    * Primary ICU admitting diagnosis of acute myocardial infarction (MI).
21. Have relative contraindications to taking TXA or have a believed adverse risk/benefit ratio for taking the drug. These include patients with:

    * Known sensitivity to TXA;
    * Recent craniotomy (past 28 days);
    * Active cerebrovascular bleed;
    * Active thromboembolic disease, (such as deep vein thrombosis, pulmonary embolism [PE], cerebral thrombosis, ischemic stroke, or acute coronary syndrome [ACS]);
    * Acute promyelocytic leukemia taking all-trans retinoic acid for remission induction or;
    * Continuing use of a combined hormonal contraceptive (including combined hormonal pill, patch or vaginal ring).
22. Exclusion for any other condition that, in the opinion of the investigator or coordinating center, would preclude the subject from being an appropriate candidate for the study.
23. Received any other investigational therapy or device within 4 weeks prior to Screening.
24. Female patients of childbearing potential with a positive urine or serum pregnancy test or who are not taking (or not willing to take) acceptable birth control measures (abstinence, intrauterine devices, contraceptive implants or barrier methods) through Day 28. Additionally, those women who are lactating and insist on breast feeding within 5 days of the last dose of study drug if their sepsis resolves.

Note: post-partum patients who have a persistent positive pregnancy test (human chorionic gonadotropin [HCG] values which have not had time to decrease) will be allowed in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-04; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tom Hallam, PhD, Study Chair — Vice President
Locations (34):
- United States (26):
  - Providence Hospital, Mobile, Alabama
  - Community Regional Medical Center, Fresno, Fresno, California
  - Long Beach Memorial Medical Center, Long Beach, California
  - UC Davis Medical Center, Sacramento, California
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - ARH Regional Medical Center, Hazard, Kentucky
  - University of Louisville Hospital Laboratory, Louisville, Kentucky
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Michigan Health Center, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic Labs - Rochester Campus, Rochester, Minnesota
  - Barnes Jewish Hospital, St Louis, Missouri
  - St. Patrick Hospital, Missoula, Montana
  - Cooper University Hospital, Camden, New Jersey
  - New York Methodist Hospital, Brooklyn, New York
  - UNC Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Mercy St. Vincent Medical Center, Clinical Research Offices, Toledo, Ohio
  - OU Medical Center, Oklahoma City, Oklahoma
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Ben Taub Hospital, Houston, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Froedtert Hospital and Medial College of Wisconsin, Milwaukee, Wisconsin
- Canada (8):
  - Peter Lougheed Centre, Calgary, Alberta
  - Foothills Medical Centre, Calgary, Alberta
  - St. Paul's Hospital, Vancouver, British Columbia
  - Royal Jubilee Hospital, Victoria, British Columbia
  - Victoria General Hospital, Victoria, British Columbia
  - St Boniface Hospital, Winnipeg, Manitoba
  - WHRA Winnipeg Health Sciences, Winnipeg, Manitoba
  - Nova Scotia Health Authority, Halifax, Nova Scotia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study from 6 sites in the US and Canada from 22 January 2015 to 18 March 2016 (day FDA was informed of decision to terminate the study).
Pre-assignment Details: The Sponsor decided to terminate this study due to slow enrollment. Throughout the study, the Sponsor made 4 protocol amendments in an effort to expand the inclusion and relax the exclusion criteria to accelerate patient enrollment. However, study was terminated after enrolling only 8 patients.
Groups:
- Tranexemic Acid: Daily a total of 700 mL of LB1148 solution containing 7.5 g of tranexemic acid will be administered orally or via NG/OG/NJ/ND/PEG tube
  LB1148
- Placebo: Daily a total of 700 mL of Placebo solution will be administered orally or via NG/OG/NJ/ND/PEG tube
  Placebo
Period: Overall Study
Arm/Group | Tranexemic Acid | Placebo
Started | 5 | 3
Completed | 5 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized subjects. The study enrolled patients with septic shock presenting with at least 1 failed organ; the sequential organ failure assessment score (SOFA score) is used to score the extent of a subjects organ failure. Enrollment allowed SOFA scores of 6-18 and trial design was stratified on baseline SOFA scores.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tranexemic Acid | Placebo | Total
Number analyzed (Participants) | 5 | 3 | 8
Age, Categorical [Count of Participants; unit: Participants] — Population: Age not collected for one patient.
  Participants
    number analyzed (Participants) | 4 | 3 | 7
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 3 | 1 | 4
    >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.59 (13.75) | 63.75 (2.26) | 56.23 (12.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 5 | 2 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 3 | 1 | 4
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 3 | 1 | 4
  United States | 2 | 2 | 4
Weight [Mean (Standard Deviation); unit: kg] | 82.76 (21.11) | 80.67 (13.96) | 81.98 (17.65)
Height [Mean (Standard Deviation); unit: cm] | 169 (13.49) | 157 (6.08) | 164.5 (12.38)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.96 (7.21) | 32.54 (3.45) | 30.30 (6.05)
SOFA Distribution at Screening [Number; unit: units on a scale] — SOFA (sequential organ failure assessment) is a morbidity severity score and mortality assessment tool focused on organ dysfunction and morbidity. The score is composed of 6 variables representing different organ systems (cardiovascular, coagulation, liver, neurological, renal and respiratory). The total score ranges from 0 to 24 with each variable having a point value range of 0 (normal) to 4 (high degree of dysfunction or failure). Since this system uses scoring of individual organ systems, it is able to measure either individual or combined organ dysfunction.
  units on a scale
    Highest Score = 6-8 | 0 | 1 | 1
    Highest Score = 9-11 | 3 | 2 | 5
    Highest Score = 12-14 | 2 | 0 | 2
    Highest Score = 15-18 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Days Alive Without Cardiovascular, Renal or Pulmonary Organ Support
Description: The patient will be classified as having organ support if organ support is required through the use of:
  * Mechanical ventilation;
  * Vasopressors to maintain adequate blood pressure (BP), or
  * Renal replacement therapy.
Time Frame: Through day 28.
Population: 5 subjects were treated with LB1148, and 3 subjects were treated with placebo. Upon review of patient charts after the study was terminated, 1 patient on placebo was enrolled on the basis of a Glasgow Coma Score calculated while under sedation, which allowed SOFA score to meet study criteria and the patient to be inappropriately enrolled.
Measure: Mean (Full Range); unit: days
Arm/Group | Tranexemic Acid | Placebo
Number analyzed (Participants) | 5 | 3
days | 14 [0 to 23] | 26 [26 to 27]

ADVERSE EVENTS:
Arm/Group | Tranexemic Acid | Placebo
Serious Adverse Events (participants affected / at risk) | 3/5 | 1/3
Other Adverse Events (participants affected / at risk) | 3/5 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tranexemic Acid (N=5) | Placebo (N=3)
Worsening Gangrene (Infections and infestations) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 1 (2) | 0 (0)
Malnutrition Status Post Dobhoff feeding tube removal (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Refractory Septic Shock (Death) (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tranexemic Acid (N=5) | Placebo (N=3)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Difficulty Swallowing (Gastrointestinal disorders) | 0 (0) | 1 (1)
Elevated AST (Investigations) | 1 (1) | 0 (0)
Fluid Overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fungal skin rash (groin and scrotum) (Infections and infestations) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypothermia (General disorders) | 1 (1) | 0 (0)
Increase in total bilirubin above lab range for normal (Investigations) | 0 (0) | 1 (1)
Left Wrist Abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Loose Stool (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pedal Edema (General disorders) | 1 (1) | 0 (0)
Possible ileus with distention and hypoactive bowel sounds (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pressure Ulcer Left Buttock (General disorders) | 1 (1) | 0 (0)
Right Hand Redness (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
SVT (15 beat run) (Cardiac disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Ventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Worsening Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Worsening Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Worsening Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to the Sponsor decision to terminate the study, data was not monitored or cleaned. The study data that are available for the 8 enrolled patients has been evaluated. However, there are too few patients to draw any meaningful conclusions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes